CLINICAL TRIAL: NCT06337032
Title: An Open-label, Single-arm Study to Provide Continued Access to Study Drug to Participants Who Have Completed Pediatric Clinical Studies Involving Gilead HIV Treatments
Brief Title: A Study to Provide Continued Access to Study Drug to Children and Adolescents Who Have Completed Clinical Studies Involving Gilead HIV Treatments
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Gilead Sciences (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: GS-US-380-6684
Record Dates: First submitted 2024-03-22; First posted 2024-03-29 (Actual); Last update posted 2025-11-05 (Actual); Status verified 2025-11

CONDITIONS: HIV-1-infection
MeSH Terms: interventions — Tablets; emtricitabine tenofovir alafenamide; Elvitegravir, Cobicistat, Emtricitabine, Tenofovir Disoproxil Fumarate Drug Combination; Cobicistat; bictegravir, emtricitabine, tenofovir alafenamide, drug combination; Ritonavir

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (4):
- Rollover from Parent Study: GS-US-311-1269: Parent Study Drug (F/TAF) or B/F/TAF (Experimental): Participants will continue to take the study drug they were taking in the parent study, emtricitabine/tenofovir alafenamide (F/TAF) along with a 3rd antiretroviral (ARV) agent. The dose of F/TAF will be based on the weight of the participant, ranging between 120/15 mg to 200/25 mg. The dose of F/TAF will be different when given with the boosted and the unboosted 3rd ARV agent: F/TAF (High Dose Tablet) for unboosted 3rd ARV agent; F/TAF (Low Dose Tablet) for the boosted 3rd ARV agent.
  Participants may switch to B/F/TAF, at a dose based on participant's weight.
  Interventions: Drug: F/TAF (High Dose Tablet); Drug: F/TAF (Low Dose Tablet); Drug: F/TAF (Lowest Dose Tablet); Drug: B/F/TAF (High Dose); Drug: B/F/TAF (Low Dose); Drug: B/F/TAF (High Dose TOS); Drug: 3rd ARV Agent
- Rollover from Parent Study: GS-US-292-0106: Parent Study Drug (E/C/F/TAF) or B/F/TAF (Experimental): Participants will continue to take the study drug they were taking in the parent study, elvitegravir/cobicistat/emtricitabine/tenofovir alafenamide (E/C/F/TAF). The dose of E/C/F/TAF will be based on the weight of the participant, ranging between 90/90/120/6 mg to 150/150/200/10 mg.
  Participants may switch to B/F/TAF at a dose based on participant's weight.
  Interventions: Drug: E/C/F/TAF; Drug: E/C/F/TAF (Low Dose); Drug: B/F/TAF (High Dose); Drug: B/F/TAF (Low Dose)
- Rollover Parent Study GS-US-216-0128: Parent Study Drug (Combination Drugs) or B/F/TAF (Experimental): Participants will continue to take the following study drugs they were taking in the parent study:
  * Cobicistat (COBI) + DRV + NRTI backbone
  * COBI + ATV + NRTI backbone
  * F/TAF + DRV+ COBI
  * F/TAF + ATV+ COBI
  * F/TAF + LPV/r
  * F/TAF + 3rd unboosted agent
  The dose of F/TAF will be based on the weight of the participant, ranging between 15/1.88 mg and 200/25 mg, once daily. Additionally, the dose of COBI will be based on the weight of the participant, ranging between 30 mg and 150 mg, once or twice daily.
  Participants may switch to B/F/TAF at a dose based on participant's weight.
  Interventions: Drug: F/TAF (High Dose Tablet); Drug: F/TAF (Lowest Dose Tablet); Drug: F/TAF (High Dose TOS); Drug: F/TAF (Low Dose TOS); Drug: F/TAF (Lowest Dose TOS); Drug: Cobicistat (High Dose); Drug: Cobicistat (Low Dose); Drug: Cobicistat (TOS); Drug: B/F/TAF (High Dose); Drug: B/F/TAF (Low Dose); Drug: B/F/TAF (High Dose TOS); Drug: B/F/TAF (Low Dose TOS); Drug: B/F/TAF (Lowest Dose TOS); Drug: 3rd ARV Agent; Drug: Nucleos(t)ide reverse transcriptase inhibitors (NRTI); Drug: ATV; Drug: DRV; Drug: Lopinavir Boosted with ritonavir (LPV/r)
- Rollover from Parent Studies: GS-US-380-1474 and CO-US-380-5578: Parent Study Drug (B/F/TAF) (Experimental): Participants will continue to take the study drug they were taking in the parent study, B/F/TAF. Participants who are diagnosed with HIV-1 infection in parent study CO-US-380-5578 and complete the study drug will continue to take the study drug they were taking in the parent study, B/F/TAF. The dose of B/F/TAF will be based on the weight of the participant.
  Interventions: Drug: B/F/TAF (High Dose); Drug: B/F/TAF (Low Dose); Drug: B/F/TAF (High Dose TOS); Drug: B/F/TAF (Low Dose TOS); Drug: B/F/TAF (Lowest Dose TOS)

INTERVENTIONS:
Drug: F/TAF (High Dose Tablet) — 200/25 mg fixed-dose combination (FDC) tablet administered orally
  Other Names: Descovy®
  Arms: Rollover Parent Study GS-US-216-0128: Parent Study Drug (Combination Drugs) or B/F/TAF; Rollover from Parent Study: GS-US-311-1269: Parent Study Drug (F/TAF) or B/F/TAF
Drug: F/TAF (Low Dose Tablet) — 200/10 mg FDC tablet administered orally
  Arms: Rollover from Parent Study: GS-US-311-1269: Parent Study Drug (F/TAF) or B/F/TAF
Drug: F/TAF (Lowest Dose Tablet) — 120/15 mg FDC tablet administered orally
  Arms: Rollover Parent Study GS-US-216-0128: Parent Study Drug (Combination Drugs) or B/F/TAF; Rollover from Parent Study: GS-US-311-1269: Parent Study Drug (F/TAF) or B/F/TAF
Drug: F/TAF (High Dose TOS) — 60/7.5 mg tablet for oral suspension (TOS) administered orally
  Arms: Rollover Parent Study GS-US-216-0128: Parent Study Drug (Combination Drugs) or B/F/TAF
Drug: F/TAF (Low Dose TOS) — 30/3.75 mg TOS administered orally
  Arms: Rollover Parent Study GS-US-216-0128: Parent Study Drug (Combination Drugs) or B/F/TAF
Drug: F/TAF (Lowest Dose TOS) — 15/1.88 mg TOS administered orally
  Arms: Rollover Parent Study GS-US-216-0128: Parent Study Drug (Combination Drugs) or B/F/TAF
Drug: E/C/F/TAF — 150/150/200/10 mg tablet administered orally
  Other Names: Genvoya®
  Arms: Rollover from Parent Study: GS-US-292-0106: Parent Study Drug (E/C/F/TAF) or B/F/TAF
Drug: E/C/F/TAF (Low Dose) — 90/90/120/6 mg tablet administered orally
  Arms: Rollover from Parent Study: GS-US-292-0106: Parent Study Drug (E/C/F/TAF) or B/F/TAF
Drug: Cobicistat (High Dose) — 150 mg tablet administered orally
  Other Names: GS-9350; Tybost®
  Arms: Rollover Parent Study GS-US-216-0128: Parent Study Drug (Combination Drugs) or B/F/TAF
Drug: Cobicistat (Low Dose) — 90 mg tablet administered orally
  Other Names: GS-9350
  Arms: Rollover Parent Study GS-US-216-0128: Parent Study Drug (Combination Drugs) or B/F/TAF
Drug: Cobicistat (TOS) — 30 mg TOS administered orally
  Other Names: GS-9350
  Arms: Rollover Parent Study GS-US-216-0128: Parent Study Drug (Combination Drugs) or B/F/TAF
Drug: B/F/TAF (High Dose) — 50/200/25 mg FDC tablet administered orally
  Other Names: Biktarvy®; GS-9883/F/TAF
Drug: B/F/TAF (Low Dose) — 30/120/15 mg FDC tablet administered orally
  Other Names: GS-9883/F/TAF
Drug: B/F/TAF (High Dose TOS) — 15/60/7.52 mg TOS administered orally
  Other Names: GS-9883/F/TAF
  Arms: Rollover Parent Study GS-US-216-0128: Parent Study Drug (Combination Drugs) or B/F/TAF; Rollover from Parent Studies: GS-US-380-1474 and CO-US-380-5578: Parent Study Drug (B/F/TAF); Rollover from Parent Study: GS-US-311-1269: Parent Study Drug (F/TAF) or B/F/TAF
Drug: B/F/TAF (Low Dose TOS) — 7.5/30/3.76 mg TOS administered orally
  Other Names: GS-9883/F/TAF
  Arms: Rollover Parent Study GS-US-216-0128: Parent Study Drug (Combination Drugs) or B/F/TAF; Rollover from Parent Studies: GS-US-380-1474 and CO-US-380-5578: Parent Study Drug (B/F/TAF)
Drug: B/F/TAF (Lowest Dose TOS) — 3.76/15/1.88 mg TOS administered orally
  Other Names: GS-9883/F/TAF
  Arms: Rollover Parent Study GS-US-216-0128: Parent Study Drug (Combination Drugs) or B/F/TAF; Rollover from Parent Studies: GS-US-380-1474 and CO-US-380-5578: Parent Study Drug (B/F/TAF)
Drug: 3rd ARV Agent — A 3rd antiretroviral (ARV) agent administered as defined by the investigator, according to the prescribing information. A 3rd ARV agent may include: boosted atazanavir (ATV), boosted lopinavir (LPV/r), boosted darunavir (DRV), unboosted efavirenz (EFV), unboosted nevirapine (NVP), unboosted raltegravir (RAL), or unboosted dolutegravir (DTG), or any other unspecified agent that is available in a participant's country
  Arms: Rollover Parent Study GS-US-216-0128: Parent Study Drug (Combination Drugs) or B/F/TAF; Rollover from Parent Study: GS-US-311-1269: Parent Study Drug (F/TAF) or B/F/TAF
Drug: Nucleos(t)ide reverse transcriptase inhibitors (NRTI) — NRTIs administered as defined by the investigator, according to the prescribing information. NRTIs may include zidovudine (ZDV), stavudine (d4T), didanosine (ddI), abacavir (ABC), tenofovir disoproxil fumarate (TDF), tenofovir alafenamide (TAF), lamivudine (3TC), or emtricitabine (FTC)
  Arms: Rollover Parent Study GS-US-216-0128: Parent Study Drug (Combination Drugs) or B/F/TAF
Drug: ATV — Administered according to the prescribing information
  Arms: Rollover Parent Study GS-US-216-0128: Parent Study Drug (Combination Drugs) or B/F/TAF
Drug: DRV — Administered according to the prescribing information
  Arms: Rollover Parent Study GS-US-216-0128: Parent Study Drug (Combination Drugs) or B/F/TAF
Drug: Lopinavir Boosted with ritonavir (LPV/r) — Administered according to the prescribing information
  Arms: Rollover Parent Study GS-US-216-0128: Parent Study Drug (Combination Drugs) or B/F/TAF

SUMMARY:
The goal of this clinical study is to provide continued access to the study drug(s) to children and adolescents with human immunodeficiency virus type 1 (HIV-1) who completed their participation in an applicable parent study and to monitor for adverse events.

The primary objectives of this study are as follows:

* To provide continued access to the study drug received in the parent protocol or switch to bictegravir/emtricitabine/tenofovir (B/F/TAF) for participants who completed a Gilead parent study evaluating drugs for HIV treatment.
* To evaluate the safety of the study drug(s) in participants with HIV-1.

ELIGIBILITY:
Key Inclusion Criteria:

* Completed an applicable parent study: GS-US-292-0106, GS-US-380-1474, GS-US-311-1269, GS-US-216-0128, or CO-US-380-5578 and gave consent to study participation.

Key Exclusion Criteria:

* Individuals planning to switch to B/F/TAF on Day 1 cannot have plasma HIV RNA ≥ 50 copies/mL during the last parent study visit prior to screening/Day 1 visit.

  * Note: individuals planning to switch after Day 1 must not have plasma HIV RNA ≥ 50 copies/mL (or detectable HIV-1 RNA level according to the local assay being used if the limit of detection is ≥ 50 copies/mL).
* Individuals planning to switch to B/F/TAF must not have any ongoing Grade 3 or 4 drug-related AE or clinically relevant Grade 3 or 4 drug-related laboratory abnormality (confirmed on repeat) related to any component of B/F/TAF prior to treatment switch.
* For those on B/F/TAF or planning to switch to B/F/TAF: previous treatment discontinuation of any component of B/F/TAF due to toxicity or intolerance.
* For those planning to switch to B/F/TAF: known hypersensitivity to any component of the study drug, its metabolites, or formulation excipients.
* Ongoing treatment with or prior use of any prohibited medications.

Note: Other protocol defined Inclusion/Exclusion criteria may apply.

Min Age: 1 Month | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 350 (Estimated)
Dates: Start 2024-08-27 (Actual); Primary Completion 2034-03 (Estimated); Study Completion 2034-03 (Estimated)

PRIMARY OUTCOMES:
Number of Eligible Participants Who Have Received Access to the Study Drug(s) in the Study | Up to 9.5 Years

SECONDARY OUTCOMES:
Percentage of Participants Experiencing Treatment-Emergent Adverse Events (TEAEs) | Up to 9.5 Years

CONTACTS AND LOCATIONS:
Overall Officials: Gilead Study Director, Study Director — Gilead Sciences
Locations (14):
- Helios Salud, Buenos Aires, Argentina
- Hospital del Niño, Panama City, Panama
- South Africa (7):
  - University of Stellenbosch, Cape Town
  - Enhancing Care Foundation, Durban
  - WITS RHI Research Centre, Johannesburg
  - Rahima Moosa Mother and Child Hospital, Johannesburg
  - Be Part Yoluntu Centre, Paarl
  - The Aurun Institute, Pretoria
  - Perinatal HIV Research Unit, Soweto
- Thailand (2):
  - Faculty of Medicine - Mahidol University, Bangkok Noi
  - Khon Kaen University, Khon Kaen
- Uganda (2):
  - Joint Clinical Research Centre, Kampala
  - Baylor College of Medicine, Kampala
- University of Zimbabwe Clinical Research Centre, Harare, Zimbabwe

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Gilead Clinical Trials Website — https://www.gileadclinicaltrials.com/study?nctid=NCT06337032